CLINICAL TRIAL: NCT06087809
Title: Improving Short Course Treatment for Common Pediatric Infections: A Randomized Quality Improvement Trial
Brief Title: Improving Short Course Treatment for Common Pediatric Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Louis Vernacchio, Director of Research, PPOC, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPOC-1
Record Dates: First submitted 2023-09-14; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Community-acquired Pneumonia; Skin Infection
MeSH Terms: conditions — Community-Acquired Pneumonia; Cellulitis | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No intervention
- Education and feedback (Experimental): Clinicians within practices assigned to the Education/Feedback group received a personal email from one of the authors at the outset of the project explaining that the Committee on Infectious Diseases of the American Academy of Pediatrics (the "Red Book Committee") recommends limiting the duration of antibiotic treatment for uncomplicated CAP to 5 days and for uncomplicated SSTI to 5-7 days. The email also shared data on the performance of the individual PCC and their practice for CAP and SSTI for the baseline period and the goals for each-50% for CAP and 67% for SST. An infographic was also attached to the email which could be printed and displayed in the PCC's work area. One month and two months into the project period, each PCC in the Education/Feedback group received an email reminding them of the recommendations and updating them on their performance since the previous email.
  Interventions: Behavioral: Education and feedback
- Clinical decision support (Experimental): Clinicians within practices assigned to the CDS group did not receive education or any performance feedback relative to the initiative. If they prescribed an antibiotic linked to a diagnosis of CAP with a duration of greater than 5 days, or to a diagnosis of SSTI with a duration greater than 7 days, they received a pop-up advisory when they attempted to sign the prescription alerting them to the relevant recommendation (eFigure 3). The alert was a "hard stop", meaning that the prescriber was required to respond in some way to continue their work. Options included altering the prescription to comply with the recommended duration or acknowledging the alert and sending the prescription with the originally selected duration.
  Interventions: Behavioral: Clinical decision support
- Combined group (Experimental): Clinicians within practices assigned to the combined group received both interventions as described above.
  Interventions: Behavioral: Education and feedback; Behavioral: Clinical decision support

INTERVENTIONS:
Behavioral: Education and feedback — Clinicians within practices assigned to the Education/Feedback group received a personal email from one of the authors at the outset of the project explaining that the Committee on Infectious Diseases of the American Academy of Pediatrics (the "Red Book Committee") recommends limiting the duration of antibiotic treatment for uncomplicated CAP to 5 days and for uncomplicated SSTI to 5-7 days. The email also shared data on the performance of the individual PCC and their practice for CAP and SSTI for the baseline period and the goals for each-50% for CAP and 67% for SST. An infographic was also attached to the email which could be printed and displayed in the PCC's work area. One month and two months into the project period, each PCC in the Education/Feedback group received an email reminding them of the recommendations and updating them on their performance since the previous email.
  Arms: Combined group; Education and feedback
Behavioral: Clinical decision support — Clinicians within practices assigned to the CDS group did not receive education or any performance feedback relative to the initiative. If they prescribed an antibiotic linked to a diagnosis of CAP with a duration of greater than 5 days, or to a diagnosis of SSTI with a duration greater than 7 days, they received a pop-up advisory when they attempted to sign the prescription alerting them to the relevant recommendation (eFigure 3). The alert was a "hard stop", meaning that the prescriber was required to respond in some way to continue their work. Options included altering the prescription to comply with the recommended duration or acknowledging the alert and sending the prescription with the originally selected duration.
  Arms: Clinical decision support; Combined group

SUMMARY:
Randomized quality improvement trial to improve the proportion of cases of community-acquired pneumonia (CAP) treated with no more than 5 days of antibiotics the proportion of cases of skin and soft tissue infections (SSTI) treated with no more than 7 days of antibiotics by primary care clinicians (PCC) within the Pediatric Physicians' Organization at Children's (PPOC), a state-wide pediatric primary care network. Interventions include education and feedback; clinical decision support (CDS) delivered at the point of care; and the combination of the two.

ELIGIBILITY:
INCLUSION CRITERIA

* Primary care clinician practicing within a PPOC primary care pediatric practice
* Treated at least one case of pneumonia or skin and soft tissue infection in calendar year 2022

EXCLUSION CRITERIA

-None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
Proportion of cases of CAP and SSTI treated with short course antibiotic treatment | 3 months
  Proportion of cases of CAP and SSTI treated with short course antibiotic treatment (<=5 days for CAP, <=7 days for SSTI)

SECONDARY OUTCOMES:
Proportion of cases of CAP treated with short course antibiotic treatment | 3 months
  Proportion of cases of CAP treated with short course antibiotic treatment (<=5 days)
Proportion of cases of SSTI treated with short course antibiotic treatment | 3 months
  Proportion of cases of SSTI treated with short course antibiotic treatment (<=7 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No